CLINICAL TRIAL: NCT05619146
Title: Upper and Lower Extremity Cycling in Incomplete Spinal Cord Injury Individuals to Promote Limb Recovery
Brief Title: Arm and Leg Cycling for Accelerated Recovery From SCI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Jose Pons, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU00216731
Record Dates: First submitted 2022-10-28; First posted 2022-11-16 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injury; Rehabilitation; Cycling
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: The participants will complete 60min of active cycling training paradigm, 5 times a week, for 12 weeks. The cycling ergometer will be used to provide motorized assistance during simultaneous arms and legs cycling to the participant while they are seated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SCI subject (Experimental): Subject with SCI
  Interventions: Device: Motor-assisted arms and legs cycling

INTERVENTIONS:
Device: Motor-assisted arms and legs cycling — The participants will complete 60min of active cycling training paradigm, 5 times a week, for 12 weeks. The cycling ergometer will be used to provide motorized assistance during simultaneous arms and legs cycling to the participant while they are seated.

SUMMARY:
The purpose of this study is to examine the ability of simultaneous motorized upper and lower extremity cycling training to regulate spinal movement patterns in order to potentially restore functional abilities (i.e., walking) in individuals with an incomplete spinal cord injury. The researchers hypothesize there will be improved walking function following motorized cycling.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) occurs at an annual rate of 50-60 per million in North America. Paralysis is also accompanied by drastic changes in independence and quality of life. SCI occurs mostly among younger individuals, half in people 16-30 years of age. Two-thirds of all SCIs are incomplete (iSCI), with some preserved neural connections relaying information to and from the brain. People with iSCI benefit most from improvements in walking. In addition to increasing independence, walking helps persons with iSCI remain active, with a variety of beneficial health-related outcomes. Therapy that can significantly increase sensorimotor function to these individuals living with iSCI for multiple decades would be hugely significant.

Currently, the most common strategies for restoring walking after an iSCI are manually intensive, including over ground walking with weight and balance support provided by multiple therapists, or with the use of expensive robotic support with controversial outcomes. Thus, the overarching goal of this proposal is to investigate if a non-specific gait rehabilitation paradigm based on motor-assisted arms and legs cycling in AIS C and D iSCI individuals generalizes to improvements in walking that outperform conventional gait specific training (Specific Aim 1). The researchers will also investigate biomechanical and motor coordination changes and adaptations tied to these functional improvements (Specific Aim 2), and the neural mechanisms that explain functional improvements and their retention over time (Specific Aim 3).

Specifically, in Specific Aim 1 the researchers will investigate the clinically-relevant gait improvements afforded by the cycling intervention. In Specific Aim 2 the researchers will focus on studying the detailed biomechanical basis for the gait improvements. In Specific Aim 3 the researchers will investigate the neuroplastic mechanisms underlying the gait improvements. For these Aims, the researchers will measure the walking gains with a battery of standard clinical tests focused on motor function, sensation, balance and spasticity (Specific Aim 1). The researchers will use motion tracking, force plates, and EMG measurement to monitor the kinematics and kinetics of gait, the neuromuscular coordination, and oxygen consumption as a measure of these energetics of walking (Specific Aim 2). In addition, the researchers will conduct a battery of physiological tests at 3-week intervals intended to detect changes in the strength of descending and ascending spinal pathways (Specific Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* Traumatic SCI T11 and above (upper motorneuron lesion)
* Incomplete paraplegia or tetraplegia (Classified as AIS C or D)
* Age range 18-75 years old, inclusive
* At least 1 year post- injury
* Independent ambulator (with normal assistive devices or bracing) for at least 10 meters (30 feet)
* Walking speed <0.8 m/s (2.62 ft/s) (or per researcher discretion)
* Bilateral arm strength to arm cycle at least 15 minutes without assistance (or per researcher discretion)

Exclusion Criteria:

* Traumatic SCI T12 and below (or lacking upper motorneuron injury)
* Complete paraplegia or tetraplegia (classified as AIS A)
* AIS B incomplete paraplegia or tetraplegia
* Presence of progressive neurologic disease
* Unable to give informed consent to participate in the study
* Significant other disease (ex: cardiological or heart disease, renal, hepatic, malignant tumors, mental or psychiatric disorders) that would prevent participants from fully engaging in study procedures
* MRI contraindications:
* Cardiac pacemaker or pacemaker wires; neurostimulators; implanted pumps
* Metal in the body (rods, plates, screws, shrapnel, dentures, metal IUD, etc)
* Surgical clips in the head or previous neurosurgery
* Cochlear implants
* Prosthetic heart valves
* Claustrophobia
* Tremor
* TMS contraindications
* Epilepsy or any other type of seizure history
* Medications that increase the risk of seizures
* Non-prescribed drug or marijuana use
* Depression, antidepressant medications, or antipsychotic medications
* Pregnancy
* Prisoners

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in 10-meter walking test (10MWT) | Changes across baseline, after 3 weeks of training, after 6 weeks of training, after 9 weeks of training, after 12 weeks of training, and 6 months after completing training.
  The 10-meter walking test (10MWT) is a physical function test measuring the total time to ambulate 10 meters in order to calculate walking speed in meters per second. A shorter time indicates a better walking speed.
Change in 6-minute walking test (6MWT) | Changes across baseline, after 3 weeks of training, after 6 weeks of training, after 9 weeks of training, after 12 weeks of training, and 6 months after completing training.
  The 6-minute walking test (6MWT) is a physical function test measuring the total distance walked in a span of six minutes will be assessed. A longer distance indicates a better walking distance.

SECONDARY OUTCOMES:
Change in motor and sensory scores (ASIA) | Changes across baseline, after 3 weeks of training, after 6 weeks of training, after 9 weeks of training, after 12 weeks of training, and 6 months after completing training.
  The American Spinal Injury Association Impairment Scale (AISA) is a standardized neurological examination used to assess the sensory and motor levels which were affected by the spinal cord injury. A clinician will assess sensory and strength in both upper and lower extremities to provide both a neurologic level of injury and classification level. The five classification levels, ranging from complete loss of neural function in the affected area (Grade A) to completely normal (Grade E). A score closer to Grade E is a better outcome.
Change in balance with the Berg balance scale (BBS) | Changes across baseline, after 3 weeks of training, after 6 weeks of training, after 9 weeks of training, after 12 weeks of training, and 6 months after completing training.
  Change in static and dynamic sitting and standing balance will be assessed using the Berg balance scale (BBS). Items are scored from zero to four. A higher score indicates better balance and decreased fall risk.
Change in walking ability with the WISCI | Changes across baseline, after 3 weeks of training, after 6 weeks of training, after 9 weeks of training, after 12 weeks of training, and 6 months after completing training.
  The Walking Index for Spinal Cord Injury (WISCI) assesses the ability of a person to walk after spinal cord injury. It consists of a rank ordering at the impairment level from most severe (0) to least severe (20) based on the amount of physical assistance required and use of assistive devices and/or braces while walking a 10-meter distance. A higher score indicates better walking ability.
Change in Modified Ashworth Scale (MAS) | Changes across baseline, after 3 weeks of training, after 6 weeks of training, after 9 weeks of training, after 12 weeks of training, and 6 months after completing training.
  The Modified Ashworth Scale (MAS) is a physical function test measuring spasticity on a 6-point ordinal scale. A score of 0 on the scale indicates no increase in tone while a score of 4 indicates rigidity. Tone is scored by passively moving the individual's limb and assessing the amount of resistance to movement felt by the examiner. A lower score is a better outcome.
Change in muscle testing or strength | Changes across baseline, after 3 weeks of training, after 6 weeks of training, after 9 weeks of training, after 12 weeks of training, and 6 months after completing training.
  Physical function test measuring strength of the muscle of interest. A muscle is isolated, and gradual external force is applied at a right angle to the muscle's long axis. Each muscle is scored on a graded scale of "weak" (score of 0) to "strong" (score of 5) based on the participant's ability to resist the external force. The test is first completed for muscles on the unimpaired side to determine normal strength before being repeated on the impaired side. Weaker participants may be tested while lying prone (gravity eliminated). A higher score value indicates higher strength and improvement.
Changes in EMG activation patterns | Changes across baseline, after 3 weeks of training, after 6 weeks of training, after 9 weeks of training, after 12 weeks of training, and 6 months after completing training.
  Electrodes will record muscle activity from the main leg muscles (e.g., soleus (SOL), tibialis anterior (TA), quadriceps (QS), hamstrings (HS)) during walking. Features closer to that of a healthy individual is a better outcome.
Changes in interlimb (upper-lower limb) modulation | Changes across baseline, after 3 weeks of training, after 6 weeks of training, after 9 weeks of training, after 12 weeks of training, and 6 months after completing training.
  This will be assessed by measuring changes in the magnitude and pattern of H-reflex suppression in the soleus (ankle extensor) of the leg during arm cycling. Features closer to that of a healthy individual is a better outcome.
Changes in the strength of cortico-spinal connectivity | Changes across baseline, after 3 weeks of training, after 6 weeks of training, after 9 weeks of training, after 12 weeks of training, and 6 months after completing training.
  This will be measured using transcranial magnetic stimulation (TMS) of the motor cortex known to produce a motor evoked potential (MEP) in the main muscles of the leg, and peak-to-peak amplitude of the MEP and recruitment curves of MEP amplitude as a function of TMS strength will be calculated and constructed. Recruitment curves closer to that of a healthy individual is a better outcome.
Changes in strength of periphery and somatosensory cortex | Changes across baseline, after 3 weeks of training, after 6 weeks of training, after 9 weeks of training, after 12 weeks of training, and 6 months after completing training.
  This will be measured using cutaneous electrodes on the arm and leg skin surface and recording the somatosensory evoked potentials (SEPs) over the primary somatosensory cortex using electroencephalography (EEG) electrodes; peak-to-peak amplitude of the SEP and recruitment curves of SEP amplitude as a function of stimulus strength will be calculated and constructed. Recruitment curves closer to that of a healthy individual is a better outcome.
Change in stride variability. | Changes across baseline, after 3 weeks of training, after 6 weeks of training, after 9 weeks of training, after 12 weeks of training, and 6 months after completing training.
  Stride variability is the ratio between the standard-deviation and mean of stride time, expressed as percentage. Decreased variability indicates a better outcome.
Change in cadence. | Changes across baseline, after 3 weeks of training, after 6 weeks of training, after 9 weeks of training, after 12 weeks of training, and 6 months after completing training.
  Cadence is the total number of steps taken within a given time period; often expressed per minute. Typically a higher number of steps is a better outcome.
Change in step length. | Changes across baseline, after 3 weeks of training, after 6 weeks of training, after 9 weeks of training, after 12 weeks of training, and 6 months after completing training.
  Step length is the distance between the point of initial contact of one foot and the point of initial contact of the opposite foot. Typically a longer step length is a better outcome, ideally with equal measurements between left and right limbs.
Change in stride length. | Changes across baseline, after 3 weeks of training, after 6 weeks of training, after 9 weeks of training, after 12 weeks of training, and 6 months after completing training.
  Stride length is the distance between successive points of initial contact of the same foot. Right and left stride lengths are normally equal. Typically a longer stride length is a better outcome, ideally with equal measurements between left and right limbs.
Change in stance time. | Changes across baseline, after 3 weeks of training, after 6 weeks of training, after 9 weeks of training, after 12 weeks of training, and 6 months after completing training.
  Stance time is the amount of time that passes during the stance phase of one extremity in a gait cycle. It includes single support and double support. Equal stance time between limbs is a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Pons, PhD, Principal Investigator — Shirley Ryan AbilityL
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No